CLINICAL TRIAL: NCT02162732
Title: Molecular-guided Therapy for the Treatment of Patients With Relapsed and Refractory Childhood Cancers
Brief Title: Molecular-Guided Therapy for Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Translational Genomics Research Institute (Other); Dell, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC009
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Neuroblastoma; Medulloblastoma; Glioma; Ependymoma; Choroid Plexus Neoplasms; Craniopharyngioma; Dysembryoplastic Neuroepithelial Tumor; Meningioma; Primitive Neuroectodermal Tumors (PNETs); Germ Cell Tumors; Rhabdomyosarcoma; Non-rhabdomyosarcoma; Ewings Sarcoma; Osteosarcoma; Wilms Tumor; Renal Cell Carcinoma; Malignant Rhabdoid Tumor; Clear Cell Sarcoma; Liver Tumors
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma; Glioma; Ependymoma; Choroid Plexus Neoplasms; Craniopharyngioma; Meningioma; Neuroectodermal Tumors, Primitive; Neoplasms, Germ Cell and Embryonal; Rhabdomyosarcoma; Sarcoma, Ewing; Osteosarcoma; Wilms Tumor; Carcinoma, Renal Cell; Rhabdoid Tumor; Sarcoma, Clear Cell; Carcinoma, Hepatocellular | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guided Therapy (Experimental): A total of 200 neuroblastoma, brain tumor, and rare tumor patients will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).
  Interventions: Device: Guided Therapy

INTERVENTIONS:
Device: Guided Therapy — A total of 200 neuroblastoma, brain tumor, and rare tumor patients will be treated. Guided therapy will allow the use of any therapeutic combination (up to 4 agents) provided it includes medications contained in the study report. All patients will be followed for survival, disease response, progression and safety. All patients will be treated according to the discretion of the treating oncologist and study committee (minimum 3 oncologists and one pharmacist). Extent of disease will be measured and assessed for changes throughout the course of the study and at 6-8 week intervals (every 2 cycles).

SUMMARY:
The purpose of this study is to test the feasibility (ability to be done) of experimental technologies to determine a tumor's molecular makeup. This technology includes a genomic report based on DNA exomes and RNA sequencing that will be used to discover new ways to understand cancers and potentially predict the best treatments for patients with cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have proven pediatric cancer with confirmation at diagnosis or at the time of recurrence/progression and clinical determination of disease for which there is no known effective curative therapy or disease that is refractory to established proven therapies fitting into one of the following categories:

   * Neuroblastoma- Patients that have relapsed following standard of care therapy (such as high risk patients, patient presenting after age 15 months or MYCN amplified, and only following (for eligible patients) high-dose chemotherapy followed by hematopoietic stem cell transplantation and maintenance therapy with retinoic acid and antibody therapy) or having progressed during standard of care therapy and non-responsive/progressive to accepted curative chemotherapy.
   * Brain Tumors
   * Medulloblastomas (At relapse after standard of care therapy [surgery, chemotherapy and/or radiation] and/or non-responsive/progressive on accepted curative therapy)
   * Gliomas (At relapse after standard of care therapy [surgery and/or radiation and/or chemotherapy] and/or non-responsive/progressive on accepted curative therapy)
   * Ependymomas (At relapse after standard of care therapy [surgery with or without radiation] and/or non-responsive/progressive on accepted curative therapy)
   * Choroid plexus tumors (At relapse after standard of care therapy [surgery] and/or non-responsive/progressive on accepted curative therapy)
   * Craniopharyngiomas (At relapse after standard of care therapy [surgery or suppressive therapy] and/or non-responsive/progressive on accepted curative therapy)
   * Dysembryoplastic neuroepithelial tumors (DNETs) (At relapse after standard of care therapy [surgery] and/or non-responsive/progressive on accepted curative therapy)
   * Meningiomas (At relapse after standard of care therapy [surgery] and/or non-responsive/progressive on accepted curative therapy)
   * Primitive Neuroectodermal Tumors (PNETs) (At relapse after standard of care therapy [surgery, chemotherapy, and/or radiation] and/or non-responsive/progressive on accepted curative therapy)
   * Germ cell tumors (At relapse after standard of care therapy [surgery, and/or radiation and/or chemotherapy] and/or non-responsive/progressive on accepted curative therapy)
   * Rare Tumors:
   * Soft tissue sarcoma Rhabdomyosarcoma (At relapse after standard of care therapy [surgery, and/or radiation, chemotherapy] and/or non-responsive/progressive to accepted curative chemotherapy) Non-rhabdomyosarcoma (At relapse after standard of care therapy [surgery, and/or radiation, chemotherapy] and/or non-responsive/progressive to accepted curative chemotherapy)
   * Bone Ewings sarcoma (At relapse after standard of care therapy [surgery, and/or radiation, chemotherapy] and/or non- responsive/progressive to accepted curative chemotherapy) Osteosarcoma (At relapse after standard of care therapy [surgery, chemotherapy] and/or non- responsive/progressive to accepted curative chemotherapy)
   * Renal Wilms tumor (At relapse after standard of care therapy [surgery, and/or radiation, chemotherapy] and/or non- responsive/progressive to accepted chemotherapy) Renal cell carcinoma (At relapse after standard of care therapy [surgery, chemotherapy] and/or non- responsive/progressive to accepted curative chemotherapy) Malignant rhabdoid tumor (At diagnosis, as there is no known curative therapy) Clear Cell Sarcoma- (At relapse after standard of care therapy [radiation, chemotherapy] and/or non- responsive/progressive to accepted curative chemotherapy) Germ Cell tumors (At relapse after standard of care therapy [surgery, chemotherapy] and/or non-responsive/progressive to accepted curative chemotherapy)
   * Liver Tumors (At relapse after standard of care therapy [surgery, chemotherapy] and/or non- responsive/progressive to accepted curative chemotherapy)
2. Subjects must be age >12 months at enrollment
3. Subjects must be age ≤ 21 years at initial diagnosis
4. Subjects must have measurable disease as demonstrated by residual abnormal tissue at a primary or metastatic site (measurable on CT or MRI) at the time of biopsy; tumor must be accessible for biopsy. In addition, subjects with bone or bone marrow only disease expected to be >75% tumor are eligible to enroll.
5. Current disease state must be one for which there is currently no known effective therapy
6. Specimens will be obtained only in a non-significant risk manner and not solely for the purpose of investigational testing.
7. Lansky or Karnofsky Score must be ≥ 50
8. Subjects without bone marrow metastases must have an ANC > 750/μl to begin treatment.
9. Subjects with CNS disease must have been on a stable dose of steroids for 2 weeks prior to their biopsy and must not have progressive hydrocephalus at enrollment.
10. Adequate liver function must be demonstrated, defined as:

    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
    * ALT (SGPT) < 10 x upper limit of normal (ULN) for age
11. A negative serum pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
12. Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
13. Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

1. Subjects who have received any cytotoxic chemotherapy within the last 7 days prior to biopsy
2. Subjects who have received any radiotherapy to the primary sample site within the last 14 days (radiation may be included in treatment decision after biopsy).
3. Subjects receiving any investigational drug concurrently.
4. Subjects with uncontrolled serious infections or a life-threatening illness (unrelated to tumor)
5. Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study

Ages: 13 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (19):
- United States (18):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics on Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Sholler GLS, Bergendahl G, Lewis EC, Kraveka J, Ferguson W, Nagulapally AB, Dykema K, Brown VI, Isakoff MS, Junewick J, Mitchell D, Rawwas J, Roberts W, Eslin D, Oesterheld J, Wada RK, Pastakia D, Harrod V, Ginn K, Saab R, Bielamowicz K, Glover J, Chang E, Hanna GK, Enriquez D, Izatt T, Halperin RF, Moore A, Byron SA, Hendricks WPD, Trent JM. Molecular-guided therapy for the treatment of patients with relapsed and refractory childhood cancers: a Beat Childhood Cancer Research Consortium trial. Genome Med. 2024 Feb 12;16(1):28. doi: 10.1186/s13073-024-01297-5. PMID 38347552
- See also: Beat Childhood Cancer — https://beatcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guided Therapy
Started | 186
Completed | 168
Not Completed | 18
Not completed — Biopsy not performed. | 18

BASELINE CHARACTERISTICS:
Population: Subjects that started at least one dose of study therapy
Arm/Group | Guided Therapy
Number analyzed (Participants) | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 134
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.04 [1 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 93
  More than one race | 0
  Unknown or Not Reported | 36
Tumor Type [Count of Participants; unit: Participants]
  Neuroblastoma | 31
  CNS Tumor | 41
  Rare Tumor | 72

OUTCOME MEASURES:

1. Primary Outcome: Days to Treatment Will be Used in Order to Determine Feasibility of Using Tumor Samples to Assess Genomic Sequencing Using Predictive Modeling to Make Real-time Treatment Decisions for Children With Relapsed/Refractory Cancers.
Description: The definition of feasibility is: Enrollment onto study, genomic profile, analysis and report generation completed, tumor board held with treatment decision, treatment review completed, start of treatment, and completion of 1 cycle of therapy.
Time Frame: 2 years
Measure: Mean (Full Range); unit: Days
Groups:
- Neuroblastoma: Subjects on study with a diagnosis of Neuroblastoma
- CNS Tumors: Subjects on study with a diagnosis of a CNS Tumor which included, but was not limited to, Ependymoma, Glioblastoma, Diffuse Midline Glioma, and Other CNS Tumors.
- Rare Tumors: Subjects on study with a diagnosis of a rare solid tumor which included, but was not limited to, Rhabdomyosarcoma, Ewing Sarcoma, Osteosarcoma, and Other Rare Tumors.
Arm/Group | Neuroblastoma | CNS Tumors | Rare Tumors
Number analyzed (Participants) | 31 | 41 | 72
Days | 31 [18 to 75] | 48 [18 to 146] | 35 [20 to 98]

2. Secondary Outcome: Number of Participants With an Unexpected Adverse Events as a Measure of Safety
Description: To determine the safety of allowing a molecular tumor board to determine individualized treatment plans
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average of 4 years.
Population: All subjects that received at least one dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Therapy
Number analyzed (Participants) | 144
Participants | 6

3. Secondary Outcome: Overall Response Rate (ORR) of Participants by the Presence of Radiologically Assessable Disease by Cross-sectional CT or MRI Imaging and/or by MIBG or PET Scans.
Description: To determine the activity of treatments chosen based on Overall response rate (ORR) using RESIST criteria. The assessment of response will include the initial measurable targets and will be performed after cycle 2, then after every other cycle. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI imaging and/or by MIBG or PET scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, At least a 20% increase in the sum of the disease measurements for measurable lesions, Stable Disease, Neither sufficient decrease to qualify for PR or sufficient increase to qualify for PD from study entry. Overall Response (OR) = CR + PR.
Time Frame: Followed until off therapy, generally 4 years
Population: Having at least one disease evaluation following completion of at least one cycle of molecular-guided therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroblastoma | CNS Tumors | Rare Tumors
Number analyzed (Participants) | 27 | 37 | 60
Participants
  Complete Response | 4 | 2 | 5
  No Evidence of Disease | 1 | 11 | 6
  Partial Response | 0 | 4 | 7
  Stable Disease | 13 | 10 | 18
  Progressive Disease | 9 | 10 | 24

4. Secondary Outcome: Progression Free Survival (PFS) Interval Will be Measured by Days and Compared to the PFS of Previous Chemotherapy Regimens Since Relapse for Each Patient.
Description: Time to progression (PFS), defined as the period from the start of the treatment until the criteria for progression are met taking as reference the screening measurements. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment (nadir), and minimum 5 mm increase over the nadir or the appearance of one or more new lesions or appearance of positive bone marrow.
Time Frame: From date of start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
Population: Time on study was measured in days from the date of initial biopsy to date of last administration of study therapy. For subjects with >1 biopsies and >1 MGT regimens, the off-therapy date from their last treatment was used.
Measure: Mean (Full Range); unit: Days
Arm/Group | Neuroblastoma | CNS Tumors | Rare Tumors
Number analyzed (Participants) | 27 | 37 | 60
Days | 153 [45 to 556] | 283 [50 to 1415] | 163 [28 to 1317]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average of 4 years.
Arm/Group | Guided Therapy
All-Cause Mortality (participants affected / at risk) | 3/144
Serious Adverse Events (participants affected / at risk) | 0/144
Other Adverse Events (participants affected / at risk) | 6/144
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Therapy (N=144)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Alanine Transaminase increased (Hepatobiliary disorders) | 1 (1)
Aspartate Transferase (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Oral Mucositis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02162732/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02162732/ICF_001.pdf